CLINICAL TRIAL: NCT07175636
Title: A Multicenter, Prospective, Phase II Clinical Trial of Short-Course Radiotherapy Followed by QL1706 Plus mFOLFOX6 as Total Neoadjuvant Therapy for Patients With pMMR/MSS Locally Advanced Rectal Cancer
Brief Title: QL1706 With Short-Course Radiotherapy and Chemotherapy for MSS Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Hai Lu, Prof, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-431
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Rectal Cancer (LARC); Mismatch Repair-Proficient (pMMR) Rectal Cancer; Non-metastatic Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short-Course Radiotherapy Followed by QL1706 Plus mFOLFOX6 (Experimental): Participants will receive short-course radiotherapy (SCRT, 25 Gy in 5 fractions over one week) followed by total neoadjuvant therapy (TNT) consisting of QL1706 (a bifunctional MabPair antibody targeting PD-1 and CTLA-4, investigational code name only) in combination with mFOLFOX6 chemotherapy for several cycles. After completion of neoadjuvant therapy, patients will undergo total mesorectal excision (TME) when operable, or may be managed with a watch-and-wait strategy if a strict clinical complete response (cCR) is achieved per institutional criteria. Standard perioperative care and follow-up will be provided.
  Interventions: Drug: Drug: QL1706 Drug: mFOLFOX6 Radiation: Short-Course Radiotherapy (SCRT)

INTERVENTIONS:
Drug: Drug: QL1706 Drug: mFOLFOX6 Radiation: Short-Course Radiotherapy (SCRT) — QL1706 is an investigational bifunctional MabPair antibody that simultaneously targets PD-1 (IgG4) and CTLA-4 (IgG1). It is administered intravenously according to the study protocol during the neoadjuvant chemotherapy cycles. The use of QL1706 aims to enhance antitumor immunity in the pMMR/MSS rectal cancer setting, a population typically unresponsive to immune checkpoint blockade alone.
  mFOLFOX6 is a standard oxaliplatin-based chemotherapy regimen composed of oxaliplatin, leucovorin, and 5-fluorouracil. It is administered in combination with QL1706 during the neoadjuvant phase as part of total neoadjuvant therapy (TNT). The regimen is modified to optimize tolerability while maintaining efficacy in locally advanced rectal cancer.
  Short-course radiotherapy consists of a total dose of 25 Gy delivered in 5 fractions over one week to the pelvis. This approach is designed to rapidly downstage tumors, release tumor antigens, and prime the immune microenvironment for subsequent immunotherapy

SUMMARY:
This is a multicenter, prospective, phase II study evaluating total neoadjuvant therapy (TNT) consisting of short-course radiotherapy (SCRT; 5×5 Gy) followed by QL1706 (a bifunctional MabPair antibody targeting PD-1 and CTLA-4, code name only) plus mFOLFOX6 chemotherapy in patients with locally advanced rectal cancer (LARC) with proficient mismatch repair/microsatellite-stable (pMMR/MSS) biology. Patients with pMMR/MSS disease derive limited benefit from immune checkpoint inhibition alone. Preclinical and clinical evidence suggests that SCRT and oxaliplatin-based chemotherapy can enhance antitumor immunity (e.g., antigen release, T-cell infiltration), providing a biological rationale for combining QL1706 with SCRT-primed TNT.

Eligible adults with cT3-4 and/or N+ mid-to-low rectal adenocarcinoma (without distant metastasis), confirmed pMMR/MSS, and ECOG 0-1 will receive: SCRT (total 25 Gy over 5 fractions), then several cycles of QL1706 plus mFOLFOX6 as neoadjuvant systemic therapy. Definitive total mesorectal excision (TME) is planned per multidisciplinary assessment; a watch-and-wait approach may be considered for patients achieving a stringent clinical complete response per institutional criteria. Standard perioperative care and postoperative follow-up will be performed.

Primary endpoint is pathologic complete response (pCR, ypT0N0) rate at surgery. Key secondary endpoints include: clinical complete response (cCR) rate, major pathologic response rate, R0 resection rate, tumor downstaging, radiologic response, disease-free survival (DFS), overall survival (OS), organ preservation rate (for patients managed non-operatively), surgical morbidity, and safety/tolerability (CTCAE v5.0). Exploratory endpoints include correlations between efficacy and baseline clinicopathologic features; optional translational analyses may investigate immune-inflammation markers related to response and resistance.

This trial aims to determine whether SCRT-primed QL1706 plus mFOLFOX6 TNT can improve tumor eradication and organ preservation while maintaining acceptable safety in pMMR/MSS LARC-a population with unmet need for effective immunotherapy-based strategies.

ELIGIBILITY:
Inclusion Criteria:

Age 18-75 years, male or female.

Histologically confirmed rectal adenocarcinoma.

Locally advanced disease (cT3-4 and/or N+, M0) based on pelvic MRI and/or CT.

Tumor located within 12 cm from the anal verge.

Proven microsatellite stability (MSS) or proficient mismatch repair (pMMR) status.

ECOG performance status 0-1.

Adequate organ function:

Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L

Platelet count ≥ 100 × 10⁹/L

Hemoglobin ≥ 90 g/L

ALT/AST ≤ 2.5 × ULN

Total bilirubin ≤ 1.5 × ULN

Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min

No prior pelvic radiotherapy, chemotherapy, immunotherapy, or targeted therapy for rectal cancer.

Signed written informed consent

Exclusion Criteria:

Evidence of distant metastasis.

Previous or concurrent malignant tumor (except cured basal cell carcinoma of skin or cervical carcinoma in situ).

Active autoimmune disease requiring systemic immunosuppressive therapy.

Active infection including hepatitis B, hepatitis C, HIV, or tuberculosis.

Known allergy or hypersensitivity to study drugs or excipients.

Uncontrolled cardiovascular disease (e.g., recent myocardial infarction, unstable angina, congestive heart failure, arrhythmia).

Pregnant or breastfeeding women.

Any condition judged by investigators to make the patient unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2029-09-20 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | At the time of surgery following completion of total neoadjuvant therapy (approximately 16-24 weeks after enrollment).
  The proportion of patients who achieve pathologic complete response, defined as the absence of viable tumor cells in both the resected primary rectal specimen and the resected lymph nodes (ypT0N0), as assessed by central pathology review.

SECONDARY OUTCOMES:
Clinical Complete Response (cCR) Rate | At response evaluation after neoadjuvant therapy and before surgery (approximately 12-20 weeks after enrollment).
  The proportion of patients achieving clinical complete response, defined by endoscopy, pelvic MRI, and digital rectal examination showing no evidence of residual tumor, based on institutional criteria.
Major Pathologic Response (MPR) Rate | At the time of surgery following neoadjuvant therapy.
  The proportion of patients with ≤10% residual viable tumor cells in the resected specimen.
R0 Resection Rate | At the time of surgery
  The proportion of patients who undergo curative resection with negative microscopic margins (R0).
Overall Survival (OS) | Up to 3 years after treatment.
  Time from enrollment to death from any cause.
Disease-Free Survival (DFS) | Up to 3 years after treatment.
  Time from surgery (or start of treatment for patients managed non-operatively) to first documented recurrence, progression, or death from any cause.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xiao WW, Chen G, Gao YH, Lin JZ, Wu XJ, Luo HL, Lu ZH, Wang QX, Sun R, Cai PQ, Zhu CM, Liu M, Li JB, Wang YR, Jin Y, Wang F, Luo HT, Li CL, Pan ZZ, Xu RH. Effect of neoadjuvant chemoradiotherapy with or without PD-1 antibody sintilimab in pMMR locally advanced rectal cancer: A randomized clinical trial. Cancer Cell. 2024 Sep 9;42(9):1570-1581.e4. doi: 10.1016/j.ccell.2024.07.004. Epub 2024 Aug 1. PMID 39094560
- [Background] Lin ZY, Zhang P, Chi P, Xiao Y, Xu XM, Zhang AM, Qiu XF, Wu JX, Yuan Y, Wang ZN, Qu XJ, Li X, Nie X, Yang M, Cai KL, Zhang WK, Huang Y, Sun Z, Hou ZG, Ma C, Cheng FZ, Tao KX, Zhang T. Neoadjuvant short-course radiotherapy followed by camrelizumab and chemotherapy in locally advanced rectal cancer (UNION): early outcomes of a multicenter randomized phase III trial. Ann Oncol. 2024 Oct;35(10):882-891. doi: 10.1016/j.annonc.2024.06.015. Epub 2024 Jul 2. PMID 38964714
- [Background] Fakih M, Sandhu J, Lim D, Li X, Li S, Wang C. Regorafenib, Ipilimumab, and Nivolumab for Patients With Microsatellite Stable Colorectal Cancer and Disease Progression With Prior Chemotherapy: A Phase 1 Nonrandomized Clinical Trial. JAMA Oncol. 2023 May 1;9(5):627-634. doi: 10.1001/jamaoncol.2022.7845. PMID 36892833
- [Background] Versluis JM, Long GV, Blank CU. Learning from clinical trials of neoadjuvant checkpoint blockade. Nat Med. 2020 Apr;26(4):475-484. doi: 10.1038/s41591-020-0829-0. Epub 2020 Apr 9. PMID 32273608
- [Background] Cercek A, Lumish M, Sinopoli J, Weiss J, Shia J, Lamendola-Essel M, El Dika IH, Segal N, Shcherba M, Sugarman R, Stadler Z, Yaeger R, Smith JJ, Rousseau B, Argiles G, Patel M, Desai A, Saltz LB, Widmar M, Iyer K, Zhang J, Gianino N, Crane C, Romesser PB, Pappou EP, Paty P, Garcia-Aguilar J, Gonen M, Gollub M, Weiser MR, Schalper KA, Diaz LA Jr. PD-1 Blockade in Mismatch Repair-Deficient, Locally Advanced Rectal Cancer. N Engl J Med. 2022 Jun 23;386(25):2363-2376. doi: 10.1056/NEJMoa2201445. Epub 2022 Jun 5. PMID 35660797
- [Background] Chalabi M, Fanchi LF, Dijkstra KK, Van den Berg JG, Aalbers AG, Sikorska K, Lopez-Yurda M, Grootscholten C, Beets GL, Snaebjornsson P, Maas M, Mertz M, Veninga V, Bounova G, Broeks A, Beets-Tan RG, de Wijkerslooth TR, van Lent AU, Marsman HA, Nuijten E, Kok NF, Kuiper M, Verbeek WH, Kok M, Van Leerdam ME, Schumacher TN, Voest EE, Haanen JB. Neoadjuvant immunotherapy leads to pathological responses in MMR-proficient and MMR-deficient early-stage colon cancers. Nat Med. 2020 Apr;26(4):566-576. doi: 10.1038/s41591-020-0805-8. Epub 2020 Apr 6. PMID 32251400
- [Background] Garcia-Aguilar J, Smith DD, Avila K, Bergsland EK, Chu P, Krieg RM; Timing of Rectal Cancer Response to Chemoradiation Consortium. Optimal timing of surgery after chemoradiation for advanced rectal cancer: preliminary results of a multicenter, nonrandomized phase II prospective trial. Ann Surg. 2011 Jul;254(1):97-102. doi: 10.1097/SLA.0b013e3182196e1f. PMID 21494121
- [Background] Schrag D, Weiser MR, Goodman KA, Gonen M, Hollywood E, Cercek A, Reidy-Lagunes DL, Gollub MJ, Shia J, Guillem JG, Temple LK, Paty PB, Saltz LB. Neoadjuvant chemotherapy without routine use of radiation therapy for patients with locally advanced rectal cancer: a pilot trial. J Clin Oncol. 2014 Feb 20;32(6):513-8. doi: 10.1200/JCO.2013.51.7904. Epub 2014 Jan 13. PMID 24419115
- [Background] Fernandez-Martos C, Pericay C, Aparicio J, Salud A, Safont M, Massuti B, Vera R, Escudero P, Maurel J, Marcuello E, Mengual JL, Saigi E, Estevan R, Mira M, Polo S, Hernandez A, Gallen M, Arias F, Serra J, Alonso V. Phase II, randomized study of concomitant chemoradiotherapy followed by surgery and adjuvant capecitabine plus oxaliplatin (CAPOX) compared with induction CAPOX followed by concomitant chemoradiotherapy and surgery in magnetic resonance imaging-defined, locally advanced rectal cancer: Grupo cancer de recto 3 study. J Clin Oncol. 2010 Feb 10;28(5):859-65. doi: 10.1200/JCO.2009.25.8541. Epub 2010 Jan 11. PMID 20065174
- [Background] Cercek A, Goodman KA, Hajj C, Weisberger E, Segal NH, Reidy-Lagunes DL, Stadler ZK, Wu AJ, Weiser MR, Paty PB, Guillem JG, Nash GM, Temple LK, Garcia-Aguilar J, Saltz LB. Neoadjuvant chemotherapy first, followed by chemoradiation and then surgery, in the management of locally advanced rectal cancer. J Natl Compr Canc Netw. 2014 Apr;12(4):513-9. doi: 10.6004/jnccn.2014.0056. PMID 24717570
- [Background] Bosset JF, Calais G, Mineur L, Maingon P, Stojanovic-Rundic S, Bensadoun RJ, Bardet E, Beny A, Ollier JC, Bolla M, Marchal D, Van Laethem JL, Klein V, Giralt J, Clavere P, Glanzmann C, Cellier P, Collette L; EORTC Radiation Oncology Group. Fluorouracil-based adjuvant chemotherapy after preoperative chemoradiotherapy in rectal cancer: long-term results of the EORTC 22921 randomised study. Lancet Oncol. 2014 Feb;15(2):184-90. doi: 10.1016/S1470-2045(13)70599-0. Epub 2014 Jan 17. PMID 24440473
- [Background] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Background] Pucciarelli S, Del Bianco P, Efficace F, Serpentini S, Capirci C, De Paoli A, Amato A, Cuicchi D, Nitti D. Patient-reported outcomes after neoadjuvant chemoradiotherapy for rectal cancer: a multicenter prospective observational study. Ann Surg. 2011 Jan;253(1):71-7. doi: 10.1097/SLA.0b013e3181fcb856. PMID 21135694
- [Background] Cunningham D, Atkin W, Lenz HJ, Lynch HT, Minsky B, Nordlinger B, Starling N. Colorectal cancer. Lancet. 2010 Mar 20;375(9719):1030-47. doi: 10.1016/S0140-6736(10)60353-4. PMID 20304247
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946